CLINICAL TRIAL: NCT07294222
Title: Establishment of Appropriate Intervention Methods for Preventing Myopia and Multimorbidity in Children and Conducting a RCT Study
Brief Title: Intervention for Preventing Myopia and Multimorbidity in Children
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Fangbiao Tao (Other)
Responsible Party: Sponsor-Investigator, Fangbiao Tao, Director of the Key Laboratory of Population Health Across Life Cycle(Anhui Medical University), Ministry of Education of the People's Republic of China, Anhui Medical University
Organization: Anhui Medical University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 81250810
Record Dates: First submitted 2025-12-07; First posted 2025-12-19 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Myopia; Mental Health; Cardiovascular Health Status
MeSH Terms: conditions — Myopia; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Usual Education Control Group (Active Comparator): Participants in this group continue with their usual school health education curriculum and do not receive the specific interventions of this study.
  Interventions: Behavioral: Standard School Health Education
- Comprehensive Lifestyle Intervention Group (Experimental): Participants in this group receive a multi-component health promotion intervention, including animated health education videos, fun health lectures, family-school environment support, and encouragement of outdoor activities using wearable devices.
  Interventions: Behavioral: Multi-component Health Promotion Package

INTERVENTIONS:
Behavioral: Standard School Health Education — Participants receive the existing health education curriculum as provided by their school, following the standard national or local guidelines, without the additional components of the study's intervention package.
  Arms: Usual Education Control Group
Behavioral: Multi-component Health Promotion Package — A 24-week program integrating: 1) Weekly animated video-based health lessons; 2) Interactive debates and handbook activities; 3) Family engagement via handbooks, meetings, and WeChat updates; 4) Health knowledge reinforcement based on fun health lectures; 5) Creation of a 'Healthy Living Corner' in classrooms; 6) Temporary use of wearable devices to monitor and encourage outdoor activity and sleep.
  Arms: Comprehensive Lifestyle Intervention Group

SUMMARY:
This study aims to develop and evaluate a scalable, hybrid intervention model for the co-prevention of myopia, obesity, and mental health issues among children. By integrating cognitive behavioral therapy principles, the model targets key modifiable lifestyle factors-including dietary nutrition, physical activity, screen time, sleep hygiene, light exposure, and psychological adaptation-through coordinated family-school engagement and online-to-offline delivery. Using a cluster randomized controlled trial design in grades 3-4 primary school students, the research will assess the effectiveness of this multi-component strategy in reducing the incidence and burden of these co-occurring conditions.

DETAILED DESCRIPTION:
This study employs a real-world, cluster randomized controlled trial (cRCT) design conducted in primary school settings. Participants will be provided with a 6-month integrated health education program involving both families and schools, accompanied by sustained environmental modifications to support healthy behaviors. Data will be collected at four time points: baseline, immediately after the intervention, 6 months, and 12 months post-baseline, to evaluate the short- and medium-term effects of the intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children in grades 3-4, aged 8-11 years.
* Informed consent obtained.

Exclusion Criteria:

* Presence of systemic diseases (e.g., endocrine, cardiac, psychiatric disorders).
* Presence of developmental abnormalities.
* Inability to complete the follow-up.

Ages: 8 Years to 11 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 4000 (Estimated)
Dates: Start 2025-12-30 (Estimated); Primary Completion 2026-12-30 (Estimated); Study Completion 2027-01-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with a Composite of Myopia, Obesity, Psychological Problems, or Cardiovascular Risk Factors at 12 Months | From enrollment to the end of treatment at 12 months

IPD SHARING:
Plan to Share IPD: No